CLINICAL TRIAL: NCT00152880
Title: Apoptosis and Hepatitis B: The Role of Apoptosis in Patients Who Are HBeAg Negative, Have Normal ALT, and HBV DNA ≥10,000 Copies/mL
Brief Title: Apoptosis and Hepatitis B: The Role of Apoptosis in Patients Who Are HBeAg Negative
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: 05-0337-T
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2005-12-01 (Estimated); Status verified 2005-09

CONDITIONS: Hepatitis B
Keywords: Hepatitis B, apoptosis
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
A large number hepatitis B surface antigen positive individuals are HBeAg negative with normal liver tests. Historically, such patients were thought to have suppressed viral replication and were considered to be at low risk for complications. With the use of more sensitive technology, physicians are now able to identify a group of patients who are HBeAg negative, have normal liver enzymes, and detectable HBV DNA. Some of these patients develop signs of liver inflammation and fibrosis on biopsy. We intend to investigate whether normal, programmed cell death (apoptosis) plays a role in causing the silent liver injury in this group of patients. In other words the purpose of this study is to see whether apoptosis may be responsible for the silent liver death and injury that occurs in these so called inactive carriers who are HBeAg negative, have normal serum ALT values and HBV DNA > 10,000 copies/mL. In this study the liver biopsies would be routinely collected in the clinic and investigated for the evidence of inflammation and fibrosis, and special testing would be performed to detect for evidence of apoptosis. Around 30 patients from UHN would be participating in this study. This study will test the hypothesis that subjects who are HBeAg negative, have normal ALT and have HBV DNA ≥10,000 copies/mL will demonstrate an increased rate of apoptosis in liver tissue compared to healthy age-matched controls. If this hypothesis is confirmed, it will imply that the previous assumption that this group of patients has inactive disease is false and would implicate apoptosis as an important mechanism responsible for causing liver damage. If apoptotic activity is indeed elevated, further study of these pathways could potentially yield therapeutic interventions to inhibit apoptosis.

DETAILED DESCRIPTION:
Through a retrospective chart review, patients with HBsAg who are HBeAg negative, have normal ALT, and HBV DNA >10,000 copies/mL and who have or who are about to undergo liver biopsy will be identified. These individuals will be patients at the Toronto Western Hospital Liver Clinics. Inclusion criteria:(1) HBsAg positive.(2) Stable HBeAg status for at least one year prior to biopsy.(3) Normal ALT levels (defined as <1.5 x the upper limit of normal) for at least 90 days prior to biopsy.(4) HBV DNA ≥10,000 copies/mL by PCR measured within 90 days of liver biopsy.Exclusion criteria:(1) Coinfection with viral hepatitis A, C or D.(2) Coinfection with HIV.(3) Presence of Hepatoma.(4) Known presence of other malignancy.(5) Previous antiviral treatment.The diagnosis of hepatitis B will be based on standard serological assay results and HBV DNA detected with polymerase chain reaction using the Cobas Amplicor HBV Monitor Test (Roche Diagnostics inc.). This testing is part of the usual blood work regularly performed on these patients.We intend to stain the liver biopsies for quantitative assessment of apoptotic activity using three staining techniques:(1) TUNEL.(2) Immunohistochemistry for activated caspase-3, caspase-9 and cytochrome-C release.(3) Western blotting for caspase 3,6,7,8 and 9. Liver biopsies will only be performed if clinically indicated independent of this study protocol.At the time of liver biopsy, liver tissue was/will be buffered in formalin and embedded in paraffin. Tissue will also be frozen at minus 80 degrees for Western blotting. Two age-matched control groups of patients will also be randomly selected and compared to the study population. These control liver biopsies will be stained for apoptotic activity and for disease activity as well. These control groups will include patients who are:(1) HBeAg negative, unstable (elevated) ALT.(2) Healthy controls (living donor biopsies). All sections will be assessed for apoptotic activity using the appropriate technique that is specific for TUNEL, immunohistochemistry and Western blotting respectively. Liver histology will also be reviewed for grade and stage by an experienced hepatopathologist at the UHN. Necroinflammatory activity will be assessed using Ishak's hepatitis activity index and the Laennec grading system (a minor modification of the METAVIR system) will be used for assessment of hepatic fibrosis. Liver cell apoptosis assessed by the various techniques will be reported for the study group and the control groups as means +/- SEM. To compare the means between groups, ANOVA or Student's t test will be performed. Pearson's correlation coefficient will be used to measure the degree of association between apoptosis and histopathological activity on liver biopsy. Only the principal investigator will have access to personal and demographic information relating to the individuals included. Those performing pathological review and statistical analysis will be blinded to patient information.

ELIGIBILITY:
Inclusion Criteria:

1. HBsAg positive.
2. Stable HBeAg status for at least one year prior to biopsy.
3. Normal ALT levels (defined as <1.5 x the upper limit of normal) for at least 90 days prior to biopsy.
4. HBV DNA ≥10,000 copies/mL by PCR measured within 90 days of liver biopsy.
5. patients attending Liver Clinic at Toronto Western Hospital, Toronto, ON, Canada

Exclusion Criteria:

1. Coinfection with viral hepatitis A, C or D.
2. Coinfection with HIV.
3. Presence of Hepatoma.
4. Known presence of other malignancy.
5. Previous antiviral treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: E.J.L (Jenny) Heathcote, MD, Principal Investigator — UHN - Toronto Western Hospital, University of Toronto
Locations (1):
- Liver Clinic, Toronto Western Hospital, UHN., Toronto, Ontario, Canada